CLINICAL TRIAL: NCT06734351
Title: A Multicenter, Evaluator and Subject-blinded, Randomized, Comparator-controlled, Parallel-design Study to Evaluate the Safety and Effectiveness of NOA VOLUME Compared to JUVÉDERM® VOLUMA® XC for Improvement of Mid-face Volume
Brief Title: A Study to Assess Safety and Effectiveness of Injections of NOA VOLUME Injectable Gel in Adult Participants Compared to JUVÉDERM VOLUMA XC for Change of Mid-Face Volume
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M21-841
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Mid Face Volume Deficit
Keywords: Mid Face Volume Deficit; NOA VOLUME; JUVÉDERM® VOLUMA® XC

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Cohort 1: NOA VOLUME (Experimental): Participants will receive NOA VOLUME on Day 1 with optional touch-up treatment on Day 31 and Month 18.
  Interventions: Device: NOA VOLUME
- Cohort 1: VOLUMA XC (Experimental): Participants will receive VOLUMA XC on Day 1 with optional touch-up treatment on Day 31 and Month 18.
  Interventions: Device: VOLUMA XC
- Cohort 2: NOA VOLUME (Experimental): Participants will receive NOA VOLUME on Day 1 with optional touch-up treatment on Day 31 and at either Month 12, 15, or 18.
  Interventions: Device: NOA VOLUME
- Cohort 2: VOLUMA XC (Experimental): Participants will receive VOLUMA XC on Day 1 with optional touch-up treatment on Day 31 and at either Month 12, 15, or 18.
  Interventions: Device: VOLUMA XC

INTERVENTIONS:
Device: NOA VOLUME — Subcutaneous and/or Supraperiosteal Plane Injection
  Arms: Cohort 1: NOA VOLUME; Cohort 2: NOA VOLUME
Device: VOLUMA XC — Subcutaneous and/or Supraperiosteal Plane Injection
  Other Names: JUVÉDERM
  Arms: Cohort 1: VOLUMA XC; Cohort 2: VOLUMA XC

SUMMARY:
Facial fullness is often regarded as a characteristic feature of a youthful face. Chronic reduction of collagen, elastin, and glycosaminoglycans contribute to the facial volume loss that characterizes the aging face. Volume restoration by replacing or augmenting soft tissue is critical to successful facial rejuvenation. NOA VOLUME is a crosslinked Hyaluronic Acid (HA) gel implant formulated with lidocaine that was developed to provide a safe, minimally invasive method of improving mid-face volume deficit. The purpose of this study is to assess safety and effectiveness of NOA VOLUME in adult participants seeking improvement of mid-face volume compared to JUVÉDERM VOLUMA XC (VOLUMA XC).

NOA VOLUME is an investigational device being developed for the improvement of mid-face volume. There will be 2 cohorts in this study. In Cohort 1, participants will receive either NOA VOLUME or VOLUMA XC with a fixed follow-up period. In Cohort 2, participants will receive either NOA VOLUME or VOLUMA XC with a variable follow-up period. Around 231 adult participants seeking improvement of mid-face volume will be enrolled in the study at approximately 15 sites in the United States.

Participants will receive either NOA VOLUME or VOLUMA XC as subcutaneous and/or supraperiosteal plane injections in the cheek on Day 1. Participants will receive optional touch-up treatment at Day 31 and optional repeat treatment at Month 18 for Cohort 1 and at Month 12, 15, or 18 for Cohort 2 and will be followed up for up to 22 months.

ELIGIBILITY:
Inclusion Criteria:

* Has moderate (3), significant (4), or severe (5) mid-face volume deficit on the 5-point photonumeric MFVDS based on evaluating investigator's (EI) live assessment.
* Mid-face is amenable to achieving at least a 1-point improvement in MFVDS score with the allowed injection volume in the treating investigator's (TI) judgement.

Exclusion Criteria:

* Significant skin laxity in the midface in the opinion of the TI.
* Significant skin pigmentation disorders or discoloration in the mid-face area that would interfere with the visual assessment of the mid-face area.
* Current cutaneous inflammatory or infectious processes (e.g., acne, herpes), abscess, unhealed wound, or cancerous or precancerous lesion on the face.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving "Responder" Status Based on the Evaluating Investigator's (EI) Live Assessment of Mid-Face Volume Deficit Scale (MFVDS) | Month 6
  A "responder" is a participant with at least 1-point improvement (reduction) of mid face volume deficit using the MFVDS. MFVDS is a validated 5-point scale (1 = None/Minimal to 5 = Severe).
Number of Participants with Adverse Events (AEs) | Up to Approximately Month 22
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Change from Baseline on the Overall Score of FACE-Q Satisfaction with Cheeks | Month 6
  The FACE-Q Satisfaction with Cheeks questionnaire is a 5-point survey where 1 = Very Dissatisfied and 4 = Very Satisfied.
Percentage of Participants Achieving "Responder" Status Based on Participant's Assessments of Global Aesthetic Improvement in the Treatment Area Using Global Aesthetic Improvement Scale (GAIS) | Month 6
  A "responder" is a participant who achieves "Improved" or "Much Improved" on GAIS. GAIS is a 5-point scale used to assess global aesthetic improvement of the treatment area (2 = Much Improved to -2 = Much Worse).
Percentage of Participants Achieving "Responder" Status Based on EI's Assessments of Global Aesthetic Improvement in the Treatment Area Using the GAIS | Month 6
  A "responder" is a participant who achieves "Improved" or "Much Improved" on GAIS. GAIS is a 5-point scale used to assess global aesthetic improvement of the treatment area (2 = Much Improved, -2 = Much Worse).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (4):
- United States (4):
  - Skin Research Institute LLC /ID# 258158, Coral Gables, Florida
  - Pure Dermatology /ID# 258168, Metairie, Louisiana
  - Aesthetic Center at Woodholme /ID# 258166, Baltimore, Maryland
  - Westlake Dermatology & Cosmetic Surgery - Westlake /ID# 258156, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M21-841